CLINICAL TRIAL: NCT01617239
Title: A Phase I, Open Label, Randomized Study in Healthy Adults to Compare Safety and Immunogenicity of Different Administration Schedules of Virosomal Influenza Vaccine
Brief Title: Clinical Study for Safety and Immunogenicity Study of Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INF-V-A017; 2012-001693-28 (EudraCT Number)
Record Dates: First submitted 2012-05-10; First posted 2012-06-12 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Influenza
Keywords: Influenza; Vaccination; Virosomal influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Inflexal V

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): 1 x standard dose (0.5 mL) on Day 1, Day 29, and Day 57
  Interventions: Biological: Virosomal influenza vaccine
- Group 2 (Experimental): 1 x double standard dose (1.0 mL) on Day 1 and 1 x standard dose (0.5 mL) on Day 57.
  Interventions: Biological: Virosomal influenza vaccine
- Group 3 (Experimental): 1 x triple standard dose (1.5 mL) on Day 1
  Interventions: Biological: Virosomal influenza vaccine

INTERVENTIONS:
Biological: Virosomal influenza vaccine — Virosomal influenza vaccine with the recommended vaccine composition for season 2011-2012:
  * 15 μg HA antigen of A/California/7/2009 (H1N1)-like virus
  * 15 μg HA antigen of A/Perth/16/2009 (H3N2)-like virus
  * 15 μg HA antigen of B/Brisbane/60/2008-like virus
  Intramuscular (i.m.) administration (M. deltoideus or M. vastus lateralis)
  Other Names: Inflexal V

SUMMARY:
The goal of the study is to assess the safety and immune response after vaccination with different doses and vaccination schedules of virosomal influenza vaccine.

DETAILED DESCRIPTION:
Virosomal influenza vaccine is usually administered intramuscularly as a single 0.5 mL dose. The aim of this study is to evaluate the safety and immunogenicity of different doses and vaccination schedules. A total of 84 healthy adults aged 18-50 years will be randomized (1:1:1) into 3 treatment groups: subjects of group 1 will receive a standard dose (0.5 mL) at Days 1, 29, and 57; subjects of group 2 will receive a double dose (1.0 mL) at Day 1 and a standard dose (0.5 mL) at Day 57; subjects of group 3 will receive a triple dose (0.5 mL) at Day 1. Local and systemic solicited adverse events up to Day 4 after each vaccination will be documented. To assess the subjects' humoral and cellular immune response against homologous and heterologous virus strains, blood will be drawn from each participant at baseline (Day 1), at the 4 subsequent monthly visits (Months 1 to 4) and at Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults
* Aged ≥ 18 to ≤ 50 years on the day of enrollment
* Written informed consent
* Female subjects of childbearing potential using and willing to continue using an acceptable method of contraception unless surgically sterilized/hysterectomized or post-menopausal for more than 2 years

Exclusion Criteria:

* Acute exacerbation of bronchopulmonary infection (cough, sputum, lung findings) or other acute disease
* Body weight below 40 kg at any visit during the study
* Acute febrile illness (≥ 38.0°C)
* Known hypersensitivity to any vaccine component
* Previous history of a serious adverse reaction to influenza vaccine
* Previous vaccination with a seasonal influenza vaccine for season 2011-2012 or a virosomal formulation of seasonal influenza vaccine in any season
* History of egg protein allergy or severe atopy
* Known blood coagulation disorder
* Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of the study vaccine, including oral corticosteroids in dosages of ≥ 0.5 mg/kg/d prednisolone or equivalent (inhaled or topical steroids are allowed)
* Known immunodeficiency (incl. leukemia, HIV seropositivity) or cancer
* Known history of psychiatric diseases, particularly dementia
* Investigational medicinal product received in the past 3 months (90 days)
* Treatment with immunoglobulins or blood transfusion(s) received in the past 3 months (90 days)
* Pregnancy or lactation
* Participation in another clinical trial for the entire duration of this trial
* Employee at the investigational site or relative of the investigator
* Subjects who in the view of investigator will not comply with study procedure and/or visit requirements as per protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of local and systemic solicited adverse events | 4 days after each vaccination (day of vaccination and the followoing 3 days)

SECONDARY OUTCOMES:
Incidence of unsolicited AEs | 4 weeks after each vaccination
Humoral and cellular immune response against homologous and heterologous vaccine strains | Baseline (before vacination) and Months 1, 2, 3, 4, and 12 after vaccination
Incidence of SAEs | up to 12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Enza di Modugno, Study Director — Crucell Holland
Locations (1):
- Center for the Evaluation of Vaccination, Unit of Epidemiology and Social Medicine, University of Antwerp, Antwerp, Belgium